CLINICAL TRIAL: NCT07296341
Title: A Phase IB/II Study To Evaluate the Safety, Tolerability, and Preliminary Efficacy of HRS-4642 Combination With Other Antitumor Therapies in Patients With Solid Tumors
Brief Title: HRS-4642 Combination With Other Antitumor Therapies in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4642-206
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced or Metastatic Pancreatic Cancer With
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-4642 combination with Adebrelimab Injection, nab-paclitaxel in combination with gemcitabine (Experimental)
  Interventions: Drug: HRS-4642;Adebrelimab Injection; nab-paclitaxel; gemcitabine
- nab-paclitaxel in combination with gemcitabine (Active Comparator)
  Interventions: Drug: HRS-4642;nab-paclitaxel; gemcitabine

INTERVENTIONS:
Drug: HRS-4642;Adebrelimab Injection; nab-paclitaxel; gemcitabine — HRS-4642 combination with Adebrelimab Injection, nab-paclitaxel in combination with gemcitabine
  Arms: HRS-4642 combination with Adebrelimab Injection, nab-paclitaxel in combination with gemcitabine
Drug: HRS-4642;nab-paclitaxel; gemcitabine — nab-paclitaxel in combination with gemcitabine
  Arms: nab-paclitaxel in combination with gemcitabine

SUMMARY:
This study is a randomized, open-label, multicenter Phase II clinical trial designed to evaluate the Safety, Tolerability and Preliminary Efficacy of HRS-4642 Combination with Other Antitumor Therapies in Patients with Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-75 years old (inclusive of both ends), gender not limited when signing the informed consent form
2. ECOG performance status 0 or 1
3. Life expectancy of greater than or equal to 12 weeks.
4. Subjects with unresectable local advanced or metastatic pancreatic cancer, and pancreatic duct adenocarcinoma confirmed by histopathology
5. Provide tumor tissue blocks fixed in formalin, embedded in paraffin, or unstained tumor specimen sections, which can be archived or freshly obtained within 3 years prior to the first study treatment (fresh acquisition is preferred).
6. At least one measurable lesion is present according to the efficacy evaluation criteria for pancreatic cancer (RECIST 1.1)

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) tumor metastasis
2. Failure to recover toxicity and/or complications from previous interventions to NCI-CTCAE ≤ Level 1 or the levels specified by inclusion and exclusion criteria
3. Subjects known or suspected to have interstitial pneumonia
4. According to the common adverse reaction event evaluation criteria NCI-CTCAE v5.0, patients with ≥ grade 3 serous fluid accumulation or imaging evidence of a large amount of abdominal fluid accumulation (those who require therapeutic puncture and drainage within 2 weeks before starting the study treatment, only those with imaging showing a small amount of ascites and no clinical symptoms can be enrolled)
5. Acute or chronic pancreatitis with significant clinical significance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the date of first dose of study drug until progressive disease (PD), death, whichever occurs first, assessed up to 16 months
  PFS is defined as the time from the date of first dose of study drug to the date of the first documentation of disease progression or date of death, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 10 months following the date the last patient was randomized
  Objective response is defined as a best confirmed response of CR or PR by RECIST v1.1 as assessed by the investigator.
disease control rate (DCR) | up to 10 months following the date the last patient was randomized
  Disease Control Rate (DCR) is defined as the frequency and percentage of participants with stable disease (SD) or CR or PR.
Duration of response (DoR) | up to 10 months following the date the last patient was randomized
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause as assessed by investigator according to RECIST v1.1.
Overall survival (OS) | From study start until target OS events have occurred (approximately 20 months after last patient enrollment)
  Overall Survival (OS) is defined as the time from the date of first dose to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided